CLINICAL TRIAL: NCT05218824
Title: Collection of Head Images During Radiotherapy (CHIRP)
Brief Title: Collection of Head Images During Radiotherapy
Acronym: CHIRP
Status: Active, not recruiting | Type: Observational
Sponsor: University of Sydney (Other)
Collaborators: Western Sydney Local Health District (Other)
Responsible Party: Sponsor
Other Study IDs: IX-2021-P0-CHIRP
Record Dates: First submitted 2021-12-08; First posted 2022-02-01 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Head and Neck Neoplasms; Radiation Therapy Complication
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary objective of this observational study is to quantify the translation, rotation, and deformation of patient head positions of head and neck cancer patients over the course of a radiation therapy treatment for head and neck cancer. This objective will be achieved by comparing X-ray images collected during each treatment session with those obtained from the planning CT scan. Secondary objectives include (1) the use of the collected X-ray images to develop realistic artificial X-ray images where patient movement can be simulated and (2) to determine whether motion can be detected from individual X-ray images acquired during radiation therapy treatment.

DETAILED DESCRIPTION:
Participants will undergo their radiation therapy treatment for HNC as planned and per the routine clinical management protocol. As part of this routine treatment, multiple x-ray images will be acquired to assist in accurate positioning of the patient for their planned radiation therapy. Normally these images are stored for a few days and then discarded. This study will be collating, storing and analysing these images. These X-ray images will be paired with the corresponding pre-treatment CT scan that is routinely acquired for each patient, as well as the locations of organs of interest, such as the tumour and surrounding structures. The patient treatment plan will also be collated, as it will allow for analysis of how any motion affects the accuracy of dose delivery. The patient radiation treatment delivery record will be collected to help sort and categorise the acquired images. Information on potential confounding or interacting factors will be collected: demographic information will be collected including sex, age, tumour stage and histology.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of head and neck cancer (any stage)
* Age 18 years or greater
* Receiving radiation therapy to the head and neck with a thermoplastic immobilisation mask
* An ECOG score in the range of 0 to 2
* Any other prior or concurrent therapy allowed

Exclusion Criteria:

* People with cognitive impairment which would preclude them from providing informed consent
* People who are unable to speak and read English and for whom obtaining consent would be difficult.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants undergoing radiation therapy at Blacktown Hospital for head and neck cancer using a thermoplastic immobilisation mask
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2022-02-14 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Translational head motion between different radiation therapy treatment sessions | 8 weeks
  Translation error (mm)
Rotational head motion between different radiation therapy treatment sessions | 8 weeks
  Rotation error (degree)
Head deformation between different radiation therapy treatment sessions | 8 weeks
  Deformation error (mm)

SECONDARY OUTCOMES:
Difference in structural similarity (SSIM) indexes between artificial and real X-rays | 8 weeks
  Image quality metric: Structural Similarity (SSIM) index.
Difference in mean absolute error between artificial and real X-rays | 8 weeks
  Image quality metric: Mean Absolute Error.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Keall, PhD, Study Chair — University of Sydney
Locations (1):
- Blacktown Hospital, Blacktown, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Yes
After study completion and publication, de-identified (non-coded, non-reidentifiable) data and medical images may be shared publicly with researchers for further scientific research. This will ensure that the potential of the data acquired in this trial is maximised. This is in accordance with the NHMRC guidelines on the publication and dissemination of research, and in line with archives, e.g. the TCIA (https://www.cancerimagingarchive.net/).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After study completion and publication, indefinitely.
Access Criteria: Data stored at the university: (i) that the data is not to be published or otherwise redistributed without the express consent of the original investigator(s) and (ii) that the data is forbidden to be used for any commercial purpose and (iii) the research is approved by an accredited ethics committee.
  Data stored at an external repository: Study data that are provided to an external research data repository will be stored at and managed by the external repository. Data will only be shared with repositories whose function has been reviewed and approved by an accredited Research Integrity/Ethics Committee/Board under a Materials Transfer Agreement with the university.